CLINICAL TRIAL: NCT01252160
Title: A Multicentre, Single-Arm, Open-Label Study Of The Repeated Administration Of QUTENZA For The Treatment Of Peripheral Neuropathic Pain
Brief Title: Safety and Effectiveness of Repeated Administration of QUTENZA Patches for Treatment of Pain Caused by Nerve Damage
Acronym: STRIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E05-CL-3001; 2009-016457-18 (EudraCT Number)
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Neuralgia, Postherpetic
Keywords: Neuralgia, Postherpetic; QUTENZA
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QUTENZA (Experimental): Cutaneous patch
  Interventions: Drug: QUTENZA

INTERVENTIONS:
Drug: QUTENZA — Cutaneous patch

SUMMARY:
In this study all patients will be treated with the same medicine, the QUTENZA patch. Subjects will receive up to 6 QUTENZA patch applications over 12 months.

DETAILED DESCRIPTION:
The rationale for the current study is to evaluate the safety of repeated QUTENZA applications, including the effect of QUTENZA on sensory function in subjects diagnosed with different types of Peripheral Neuropathic Pain (PNP). In order to adequately assess the long-term safety QUTENZA in well defined patient populations the current study will enroll a minimum of 100 patients each with HIV-Associated Neuropathy (HIV-AN) and Postherpetic Neuralgia (PHN).

ELIGIBILITY:
Common Inclusion Criteria:

* Be in good health as determined by the investigator
* Average pain score >=4 during screening period (using the average reported pain from the Brief Pain Inventory [BPI])
* Intact, non-irritated, dry skin over the painful area(s) to be treated
* All females of child bearing potential must be willing to use effective methods of birth control during the study and for 30 days following study termination
* Be willing and able to comply with protocol requirements for the duration of study participation

Population-specific Inclusion Criteria:

* All subjects must meet one (and only one) of the Population-Specific Inclusion Criteria for PHN, HIV-AN, PNI or ISNN or have adequately characterized PNP based on clinical history and examination.

  * Postherpetic Neuralgia (PHN): Prior diagnosis of PHN with pain persisting at least 3 months since shingles vesicle crusting, documented by the primary treating physician or investigator
* Or

  * Painful HIV-Associated Neuropathy (HIV-AN): Presence of HIV-AN existing for a minimum of 3 months, confirmed using the Brief Peripheral Neuropathy Screen (BPNS) at the time of study entry
* Or

  * Peripheral Neuropathic Injury (PNI): Diagnosis of Post-traumatic Peripheral Neuropathic Pain syndrome, including post-surgical neuropathic pain, neuropathic pain due to peripheral nerve injury, confirmed by a qualified pain specialist and persisting for a minimum of 3 months following the traumatic event
* Or

  * Idiopathic Small Nerve Neuropathy (ISNN): Diagnosis of ISNN based on clinical criteria (e.g. quantitative sensory testing) or skin biopsy

    1. Neuropathy exclusively or predominantly affecting A-δ (small myelinated) and nociceptive C (unmyelinated) nerve fibres
    2. Loss of pinprick and temperature sensation in feet
* Or

  * Other Peripheral Neuropathic Pain (PNP): Adequately characterized PNP based on clinical history and examination existing at the time of screening

Exclusion Criteria:

* Any prior receipt of QUTENZA open label or blinded study patches
* Use of oral or transdermal opioids exceeding a total daily dose of morphine of 80 mg/day, or equivalent; or any parenteral opioids, regardless of dose, within 7 days preceding the first patch application visit
* Lack of an effective pain medication strategy for the subject, such as unwillingness to use opioid analgesics during study treatment, or high tolerance to opioids precluding the ability to relieve treatment-associated discomfort with oxycodone or other analgesic, as judged by the investigator
* Active substance abuse or history of chronic substance abuse within 1 year prior to enrolment or prior chronic substance abuse (including alcoholism) likely to re-occur during the study period as judged by the investigator
* Use of any topical pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics, steroids or capsaicin products on the painful areas within 7 days preceding the first patch application visit
* Current use of any investigational agent (excluding antiretrovirals in Phase 3 evaluation to treat HIV infection)
* Unstable or poorly controlled hypertension or a recent history of a cardiovascular event which, in the opinion of the investigator, would put the patient at risk of adverse cardiovascular reactions related to the patch application procedure
* Evidence of another contributing cause for peripheral neuropathy, and/or treatment within 90 days prior to screening visit with any drug that may have contributed to the sensory neuropathy
* Past or current history of Type I or Type II diabetes mellitus
* Current psychotic disorders
* Clinically significant abnormal ECG at screening
* Hypersensitivity to capsaicin (i.e., chilli peppers or Over-the-counter [OTC] capsaicin products), any QUTENZA excipients, local anesthetics, oxycodone, hydrocodone, or adhesives
* Significant ongoing or untreated abnormalities in cardiac, renal, hepatic, or pulmonary function that may interfere either with the ability to complete the study or the evaluation of adverse events
* Significant pain of an aetiology other than painful HIV-AN, PHN, PNI, ISNN or other adequately characterized PNP for example, compression-related neuropathies (e.g., spinal stenosis), fibromyalgia or arthritis
* Posttraumatic neuropathic pain due to Complex Regional Pain Syndrome (CRPS, Type I)
* Active malignancy or history of malignancy during the past 5 years (a history of squamous cell carcinoma or a basal cell carcinoma not involving the area to be treated is allowed)
* Evidence of cognitive impairment including dementia that may interfere with subject's ability to complete study evaluations and recall pain levels in the past 24 hours
* Planned elective surgery during the trial
* Neuropathic pain areas located only on the face, above the hairline of the scalp, and/or in proximity to mucous membranes
* Female subjects of child-bearing potential with a positive serum or urine pregnancy test prior to treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2010-10-28 (Actual); Primary Completion 2013-09-26 (Actual); Study Completion 2013-09-26 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Throughout the study up to 65 weeks
Serious adverse events (SAEs) | Throughout the study up to 65 weeks
Treatment-emergent adverse events | Throughout the study up to 65 weeks
Proportion of subjects who prematurely terminate from the study due to an AE | Throughout the study up to 65 weeks
Change in Sensory function | All visits throughout the study up to 65 weeks

SECONDARY OUTCOMES:
Use of concomitant pain medications following each patch application | Throughout the study up to 65 weeks
Change from baseline in Vital signs | All visits throughout the study up to 65 weeks
Dermal assessment score | All visits throughout the study up to 65 weeks
The proportion of subjects completing at least 90% of the intended patch application duration | All visits throughout the study up to 65 weeks
Neurological assessment | All visits throughout the study up to 65 weeks
Brief Pain Inventory (BPI) | Throughout the study up to 65 weeks
Patient Global Impression of Change (PGIC) | All visits throughout the study except the first patch application visit up to 65 weeks
European Quality of life questionnaire in 5 Dimensions (EQ5D) | All visits throughout the study except the screening visit and unscheduled visits up to 65 weeks
Hospital Anxiety and Depression Score (HADS) | All visits throughout the study except the screening visit and unscheduled visits up to 65 weeks
Work Productivity and Activity Impairment Questionnaire: Neuropathic Pain (WPAI:NP) | All visits throughout the study except the screening visit and unscheduled visits up to 65 weeks
Self-Assessment of Treatment (SAT) questionnaire | At the Week 26 visit and planned or early termination visit no later than week 65
Change in use of concomitant pain medications | Throughout the study up to 65 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe Ltd.
Locations (54):
- Vienna, Austria
- Belgium (5):
  - Antwerp
  - Brussels
  - Edegem
  - Genk
  - Roeselare
- Czechia (3):
  - Brno-Bohunice
  - Plzen-Lochotin
  - Prague
- Finland (2):
  - Helsinki
  - Tampere
- France (4):
  - Boulogne-Billancourt
  - Nice
  - Paris
  - Saint-Etienne
- Athens, Greece
- Pécs, Hungary
- Ireland (2):
  - Cork
  - Dublin
- Italy (9):
  - Chieti
  - Milan
  - Naples
  - Palermo
  - Pavia
  - Rimini
  - Rionero in Vulture
  - Roma
  - Taormina
- Netherlands (2):
  - Nieuwegein
  - Zwolle
- Poland (4):
  - Bydgoszcz
  - Katowice
  - Lodz
  - Warsaw
- Romania (2):
  - Bucharest
  - Timișoara
- Bratislava, Slovakia
- Slovenia (2):
  - Jesenice
  - Ljubljana
- Spain (9):
  - Badalona
  - Barakaldo
  - Barcelona
  - Cataluna
  - Ferrol
  - Granada
  - Madrid
  - Málaga
  - Salamanca
- United Kingdom (6):
  - Brighton
  - Edinburgh
  - Glasgow
  - Liverpool
  - London
  - Solihull

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473
- See also: Link to results on EudraCT website — https://www.clinicaltrialsregister.eu/ctr-search/trial/2009-016457-18/results
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=81